CLINICAL TRIAL: NCT03109483
Title: Effectiveness of the Geriatric Activation Program Pellenberg (GAPP) on the Geriatric Rehabilitation Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Margreet van Dijk, Physical Therapist, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S59948 / B322201731432
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Stroke; Hip Fractures; Abdominal Injury; Chronic Obstructive Pulmonary Disease
Keywords: geriatric patients; elderly; multicomponent physical therapy
MeSH Terms: conditions — Stroke; Hip Fractures; Abdominal Injuries; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: explorative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geriatric Activation Program Pellenberg (Other): intensive multicomponent physical therapy week program
  Interventions: Other: Geriatric Activation Program Pellenberg

INTERVENTIONS:
Other: Geriatric Activation Program Pellenberg — intensive multicomponent physical therapy week program

SUMMARY:
The aim of this study is to investigate the effectiveness of our developed week-treatment program GAPP, on strength, balance, speed, functionality and cognition, with the main goal to achieve a better independence for activities of daily living (ADL).

Each day of the week an exercise program of 45 minutes is given assigned to a specific aspect of the rehabilitation; strength, balance, speed, functional training and one day is for testing or group therapy.

Participants will be followed for four weeks, with testing on day one, after two weeks and at the last day of the four-week program.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness of our developed week-treatment program GAPP (Geriatric Activation Program Pellenberg), on strength, balance, speed, functionality and cognition, with the main goal to achieve a better independence for ADL.

Each day of the week an exercise program of 45 minutes is given assigned to a specific aspect of the rehabilitation.

Monday: speed and coordination, including as many repetitions as possible in one minute for: quick arm movements in standing, quick trunk movements in sitting, quick weight transfers in standing, stepping.

Tuesday: functional training, including walking stairs, transfers, sitting to lying and reverse, moving objects in the room, functional fit-o-meter.

Wednesday: balance, including maximum weight transfers in all directions, exercises with reduced base of support, reaching.

Thursday: strength, including sit to stand with a weight belt, lifting a weight bimanual of the table, walking with ankle weights, arm extension with therapy bands.

Friday: testing or group activity. One week the following test will be taken: Berg Balance Scale, 10m walking test, Digit Symbol Substitution Test, knee extension and elbow extension strength with the microfet2, Basic-ADL and Geriatric Depression Scale.

The other week there will be a group session, this could be in sitting (like moving on music) or standing (like petanque).

Walking will be practiced every day of the week and individual needs (like specific hand rehabilitation or pain problems) will be addressed besides the program when needed.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the geriatric rehabilitation ward of UZ Leuven, campus Pellenberg
* the ability to walk 10m with help of a person or walking aid
* an expected stay of at least four weeks
* a signed informed consent

Exclusion Criteria:

* medically instable
* not able to understand the questions and tasks of the program or testing

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Independence for activities of daily living | four weeks
  Independence for ADL measured with the Basic-ADL
Functional Balance | four weeks
  Functional balance measured with the Berg Balance Scale

SECONDARY OUTCOMES:
Walking speed | four weeks
  Walking speed measured with the 10m walking test
Strength of arm Extension | four weeks
  Strength of arm extension, measured with the microFET2 hand held dynamometer. The mean peak force in Newton of three trail will be used.
Strength of knee extension | four weeks
  Strength of Knee extension, measured with the microFET2 hand held dynamometer. The mean peak force in Newton of three trail will be used.
Cognitive function | four weeks
  The Digit Symbol Substitution Test will be used to measure response speed, sustained attention
General state of mind | four weeks
  General state of mind measured with the Geriatric Depression Scale 15

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaire Ziekenhuizen Leuven, campus Pellenberg, Pellenberg, Belgium

IPD SHARING:
Plan to Share IPD: No